CLINICAL TRIAL: NCT06134609
Title: Does Sexual Intercourse Affect the Outcomes of Frozen-thawed Embryo Transfer? Randomized Controlled Trial
Brief Title: Does Sexual Intercourse Affect the Outcomes of Frozen-thawed Embryo Transfer?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Dror Lifshitz, Principal Investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SMC-0653-23
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Embryo Transfer; Fertilization in Vitro; Coitus
Keywords: IVF; Embryo Transfer; Sexual intercourse; Coitus; Pregnancy
MeSH Terms: conditions — Coitus | interventions — Sex

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, clinical trial. Patients will be randomized into two groups (by concealed envelopes). The study group is subjected to have intercourse without using a condom at the evening/night after the embryo transfer, while the control group is subjected to abstain for the next 48 hours after the transfer.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned to intercourse (Experimental): The study group is subjected to perform intercourse without using a condom at the evening/night after the embryo transfer
  Interventions: Behavioral: Sexual intercourse
- Assigned to abstain (No Intervention): The control group is assigned to abstain from coitus the next 48 hours after the embryo transfer.

INTERVENTIONS:
Behavioral: Sexual intercourse — Sexual intercourse without barrier contraceptive at the evening/night after the embryo transfer
  Arms: Assigned to intercourse

SUMMARY:
The goal of this clinical trial is to test whether sexual intercourse the night after embryo transfer affects thawed embryo implantation rates. Women undergoing one of their first four frozen embryo transfers with a good quality embryo will be randomly assigned to two groups. The study group is subjected to have intercourse without using a condom at the evening/night after the embryo transfer, while the control group will abstain from intercourse for the next 48 hours after the transfer. Researchers will compare the ongoing pregnancy rates between the intervention group and the control group.

DETAILED DESCRIPTION:
It is currently unclear whether sexual intercourse the night after embryo transfer, with or without semen ejaculation, is detrimental to thawed embryo implantation rates.

The following study is a prospective, randomized, clinical trial, including patients attending our university-affiliated Infertility and IVF center.

The goal of this clinical trial is to test whether coitus the night after embryo transfer affects thawed embryo implantation rates. At the day of the embryo transfer women (ages 18-41yrs) undergoing one of their first four frozen embryo transfers with a good quality embryo will be randomly assigned to two groups. The study group is subjected to have intercourse without using a condom at the evening/night after the embryo transfer, while the control group is subjected to abstain for the next 48 hours after the transfer.

The day after the embryo transfer an electronic questionnaire will be sent to the patients to confirm whether they had intercourse or not. The questionnaire will also address whether male ejaculation was performed intravaginally and whether female orgasm occurred.

12-14 days after the embryo transfer a BHCG serum test will be performed. For those patients with a negative BHCG test surveillance will be stopped. For those with a positive BCHG test a gynecologic US will be performed at week 6. After wards surveillance will cease for all participants. Researchers will compare the ongoing pregnancy rates between the intervention group and the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Women age 18-41yrs.
2. BMI (body mass index) of 18-35 kg/m².
3. Patients undergoing one of their first four frozen embryo transfers.
4. Patients transferring a good quality embryo, either a cleavage stage embryo or a day 5 blastocyst.

Exclusion Criteria:

1. Patients age above 42.
2. Moderate or poor-quality embryos.
3. Patients with hydrosalpinx or uterus malformations.
4. Patients who are not able or are not interested in having vaginal intercourse (same sex couples for example).
5. Couples undergoing preimplantation genetic diagnosis when natural cycle frozen embryo transfer is planned (as they are instructed to avoid intercourse).

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 656 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | At 6 week of gestation (4 weeks after embryo transfer)
  Ultrasound showing a fetus with a heartbeat

SECONDARY OUTCOMES:
Biochemical pregnancy rate | 12-14 days after the embryo transfer
  Positive BHCG blood test
Clinical pregnancy rate | At 6 week of gestation (4 weeks after embryo transfer)
  Ultrasound confirmation of an intrauterine gestational sac

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crawford G, Ray A, Gudi A, Shah A, Homburg R. The role of seminal plasma for improved outcomes during in vitro fertilization treatment: review of the literature and meta-analysis. Hum Reprod Update. 2015 Mar-Apr;21(2):275-84. doi: 10.1093/humupd/dmu052. Epub 2014 Oct 3. PMID 25281684
- [Background] Robertson SA, Sharkey DJ. Seminal fluid and fertility in women. Fertil Steril. 2016 Sep 1;106(3):511-9. doi: 10.1016/j.fertnstert.2016.07.1101. Epub 2016 Jul 30. PMID 27485480
- [Background] Fanchin R, Righini C, Olivennes F, Taylor S, de Ziegler D, Frydman R. Uterine contractions at the time of embryo transfer alter pregnancy rates after in-vitro fertilization. Hum Reprod. 1998 Jul;13(7):1968-74. doi: 10.1093/humrep/13.7.1968. PMID 9740459
- [Background] Saccone G, Di Spiezio Sardo A, Ciardulli A, Caissutti C, Spinelli M, Surbek D, von Wolff M. Effectiveness of seminal plasma in in vitro fertilisation treatment: a systematic review and meta-analysis. BJOG. 2019 Jan;126(2):220-225. doi: 10.1111/1471-0528.15004. Epub 2017 Dec 6. PMID 29078039
- [Background] Hou JW, Yuan LH, Cao XL, Song JY, Sun ZG. Impact of sexual intercourse on frozen-thawed embryo transfer outcomes: a randomized controlled trial. Contracept Reprod Med. 2023 Mar 2;8(1):19. doi: 10.1186/s40834-023-00218-y. PMID 36859338